CLINICAL TRIAL: NCT07246590
Title: COVE-2: A Phase 3, Double-blind, Randomized, Vehicle-controlled Study to Evaluate the Efficacy and Safety of YCANTH (VP-102) in Subjects With Common Warts (Verruca Vulgaris)
Brief Title: Cantharidin Application in Patients With Common Warts (Verruca Vulgaris) (COVE-2)
Acronym: COVE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Verrica Pharmaceuticals Inc. (Industry)
Collaborators: Canfield Scientific Inc. (Unknown); Medidata Solutions (Industry); Veeva Systems (Industry); Torii Pharmaceutical Co. Ltd. (Unknown); Allucent (US) LLC (Unknown); Myonex LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-CW-301
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Common Warts; Common Warts (Verruca Vulgaris); Human Papilloma Virus (HPV); Warts
Keywords: Common Warts; Common Warts (Verruca Vulgaris); Human Papilloma Virus (HPV)
MeSH Terms: conditions — Warts | interventions — VP-102

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VP-102 (Experimental): Topical solution, which is a light violet to dark purple, slightly viscous liquid.
  0.7% (each mL contains 7 mg of cantharidin)/glass ampule within an applicator. Each applicator contains 0.45 mL of 0.7% w/v cantharidin. Administered Topical/every 21 (± 4) days. All treatments will take place within a 75-day period.
  Interventions: Combination Product: VP-102
- Vehicle (Placebo Comparator): Topical solution, which is a light violet to dark purple, slightly viscous liquid.
  No active drug/glass ampule within an applicator. Each applicator contains 0.45 mL of 0.7% w/v cantharidin. Administered Topical/every 21 (± 4) days. All treatments will take place within a 75-day period.
  Interventions: Combination Product: Vehicle

INTERVENTIONS:
Combination Product: VP-102 — A single-use applicator and applied in sufficient quantity to cover the entirety of each treatable common wart, including approximately a 1 to 2 mm margin of surrounding, healthy skin. The contents of no more than 2 applicators may be applied at each treatment visit. Each applicator contains 0.45 mL of 0.7% w/v cantharidin.
  Occlusive tape (occlusive tape with similar properties should be used across all clinical sites) will be applied to warts that have been treated. Once applied, the occlusive tape should be gently rubbed to maximize adherence to the treated area.
  Arms: VP-102
Combination Product: Vehicle — Vehicle is contained in a single-use applicator and applied in sufficient quantity to cover the entirety of each treatable common wart, including approximately a 1 to 2 mm margin of surrounding, healthy skin. The contents of no more than 2 applicators may be applied at each treatment visit. The Vehicle applicator contains the same excipient formulation as the VP-102 applicator but does not contain the active pharmaceutical ingredient cantharidin.
  Occlusive tape (occlusive tape with similar properties should be used across all clinical sites) will be applied to warts that have been treated. Once applied, the occlusive tape should be gently rubbed to maximize adherence to the treated area.
  Arms: Vehicle

SUMMARY:
This is a Phase 3, double-blind, randomized, vehicle-controlled study (Study number VP-CW-301; referred to as COVE-2 [Cantharidin and Occlusion in Verruca Epithelium]) to evaluate the efficacy and safety of YCANTH (VP-102) treatment in subjects with common warts.

DETAILED DESCRIPTION:
Methodology:

This Phase 3, double-blind, randomized, vehicle-controlled study (Study number VP-CW-301; referred to as COVE-2 [Cantharidin and Occlusion in Verruca Epithelium 2]) includes a Screening Period of up to 60 days, followed by a 75-day Treatment Period, and a 63-day Follow-up Period.

Treatments:

Treatment Visit 1 (Day 1), the day of the first application of study drug (YCANTH [VP-102] or Vehicle), may occur on the same day as the Screening Visit. Dermatologic examination, wart measurements, location of all treatable common warts, and evaluation of response to treatment (ERT; as defined in Assessments and procedures) must be repeated if the Screening Visit and Treatment Visit 1 do not coincide. YCANTH (VP-102) or Vehicle will be applied by the Investigator or qualified member of the research team. Study drug will be applied to treatable common warts, including an approximate 1 to 2 mm margin of healthy, surrounding skin. Warts are to be treated, then covered with occlusive tape (occlusive tape with similar properties should be used across all clinical sites) that will remain in place overnight and be removed just before the 24 hour evaluation of response to treatment (ERT).

Before application of study drug, wart paring, if necessary, will be completed. If adherent scale is not present, study drug can be applied without paring.

Treatment will continue every 21 (±4) days until complete clearance of all warts or a maximum of 4 treatment sessions during the 75-day treatment period. The exact treatment interval will be determined by evaluation of the treatment site, taking into account ongoing local skin reactions (LSRs), which are defined as temporary local skin reactions (vesiculation, pain, pruritus, scabbing, erythema, discoloration, application site dryness, edema and erosion. that are expected and consistent with historical treatment with YCANTH (VP-102). Subjects will be required to return for every treatment and follow-up visit even if their treatable common warts have cleared. Subjects will have an in- person visit 24 (± 6) hours after Treatment Visit 1 (first application of study drug). After Treatment Visits 2, 3, and 4 (Days 21, 42, and 63, respectively), telephone follow-up will be conducted 24 to 72 hours after application of study drug. In addition, telephone follow-up will be conducted 7 to10 days after application of study drug after Treatment Visits 1,2,3 and 4. During the telephone calls, a member of the research team will complete ERT assessments and inquire about AEs and concomitant medications.

Assessment for complete clearance (i.e., complete resolution of all common warts as assessed visually by a Blinded Assessor) may be made once all treatable common warts are evaluable and not obscured by an ongoing LSR. If the Investigator is unable to evaluate or treat 1 or more warts due to ongoing LSRs, no warts should be treated; the visit will be documented as an Unscheduled Visit. The timing of the next visit will be determined by resolution of the LSRs. All LSRs must resolve sufficiently to allow for evaluation of the treatment site. The research team will be in contact with the subject until all LSRs are resolved. Once LSRs have resolved, a Treatment Visit will be scheduled within 21 (± 4) days of the previous treatment application, noting it may be longer than 21 (± 4) days depending on the length of time until LSR resolution. A treatment interval exceeding 21 (± 4) days because of resolving LSRs will not be considered a protocol deviation.

All treatable common warts that are not completely clear should undergo treatment with study drug. No partial treatment of treatable common warts is permitted, unless a subject would be required to exceed the maximum number of 2 applicators per treatment session in order to complete treatment. Each applicator can cover approximately 1500 mm2 for a total of approximately 3000 mm2 using the 2 study drug applicators.

If a subject receives fewer than 4 treatments within the 75-day treatment period because of the duration of post-treatment LSRs, this will not be considered a protocol deviation. No treatment should be administered after the 75-day treatment period without Sponsor approval.

Subjects will be required to attend all visits even if they have achieved complete clearance of all treatable common warts at a previous visit.

Subjects enrolled in this study (COVE-2) will be eligible to enroll in a Long-Term Follow-up (LTFU) study (Study VP-CW-303 [COVE-4]) to evaluate the safety and efficacy of YCANTH (VP-102) over 54 weeks:

* Subjects who have completed the in-person Day 84 (0 to + 8 days; End-of-Treatment/End-of-Study 1) Visit and have complete clearance will be assessed at follow-up visits on Day 105 (± 7 days; Follow-up 1/End-of-Study 2) and Day 147 (± 7 days; Follow-up 2/End-of-Study 3).
* Subjects who have not achieved complete clearance of all treatable common warts by Day 84, and those who have new treatable common warts or recurrence of previously treated warts after Day 84 (ie, at Day 105 or Day 147) will be eligible to transition into the LTFU study.
* At Day 147, all subjects remaining in COVE-2 will be eligible to transition into the LTFU study for continued follow-up and treatment.

In the LTFU study, subjects will receive open-label YCANTH (VP-102) every 21 days until all treatable common warts are clear (for a maximum of 4 additional treatments) or until Day 357, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Candidates will be included in the study if they:

1. Are male or female patients ≥ 2 years of age.
2. Are immunocompetent.
3. Have a minimum of 1 treatable common wart (verruca vulgaris) of any size and height:

   1. Common warts are considered treatable if they are located anywhere on the body, except for the following excluded areas: the eye area (including eyelids), lips, oral cavity, nasal cavity, inside of the ears, soles of the feet (plantar warts), subungual spaces (ie, under the fingernail or toenail), or the anogenital area (warts within 10 mm of a mucosal surface should not be treated).
   2. Common warts located in excluded areas (warts within 10 mm of a mucosal surface) will not be treated or evaluated in this study. Warts that are genital, plantar, or anal are not considered common warts and are thus excluded from treatment and evaluation in this study. A subject will not be excluded from the study if they have these types of warts, but the subject must also have warts that meet the inclusion criteria.

      * If treatment of these excluded wart types is required during the study, it should be limited to destructive therapy such as cryosurgery and warts cannot be within 10 mm of any warts that are under study.
4. Have no systemic or dermatologic disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs.
5. Agree to refrain from swimming, bathing, or prolonged immersion in water or any liquids until the study drug is removed after each treatment.
6. Have the ability, or have a parent/guardian with the ability, to follow study instructions and the willingness to complete all study requirements.
7. Agree not to use any wart-removing product (prescription or over-the-counter) other than the study drug during the course of the study, with the exception of circumstances allowed under Inclusion Criterion 3b.
8. Provide written informed consent or assent in a manner approved by the IRB and/or have a parent/guardian provide written informed consent as evidenced by the signature on an IRB approved assent/consent form. Subjects who turn 18 years of age (or legal age per state or country) during the study will be required to re-consent to remain on the study.
9. Provide written authorization for use and disclosure of protected health information (per state and/or country requirements).
10. If participating in the optional photographic assessment, agree to allow photographs of treatable common warts to be taken at selected visits by the research team.

Exclusion Criteria:

Candidates will be excluded from the study if they:

1. Are unable to cooperate with the requirements or visits of the study, as determined by the Investigator.
2. Have any warts present at Baseline in an allowed anatomic location that the subject, parent/guardian, or Investigator is unwilling to treat.
3. Plantar warts and external genital warts will not be included in this study, in addition, subungual warts and warts within 10 mm of a mucosal surface will not be included in this study due to their anatomical location and complex treatment modalities.
4. Are systemically immunosuppressed or have taken required systemic immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 30 days before enrollment or such treatment is planned to be required during the course of the study. Routine use of local (eg, topical, inhaled, intranasal) corticosteroids and episodic use of systemic medications to treat conditions arising during the study is allowed.
5. Have any chronic or acute medical condition that, in the opinion of the Investigator, may interfere with the study results or place the subject at undue risk (eg, human immunodeficiency virus, systemic lupus erythematosus, viral hepatitis, uncontrolled diabetes).
6. Have had any previous treatment (including an investigational agent in a clinical trial) of common warts, including but not limited to the use of cantharidin, imiquimod, antivirals, retinoids, topical salicylic acid, lactic acid, hydrogen peroxide, trichloroacetic acid, pulse dye laser, iodine-based or nitric oxide-based therapies, oral cimetidine, coix seed, intralesional immunotherapy, curettage, or freezing of warts in the 90 days before treatment.
7. Have more common warts, or wart area, to be treated than can be adequately covered with the contents of 2 study drug applicators, as determined by total wart surface area. Each applicator can cover approximately 1500 mm2 for a total of approximately 3000 mm2 using the 2 study drug applicators.
8. Immunizations (eg, flu shots) may be administered throughout the study, but not within 5 days before or after any treatment with study drug and will be recorded as concomitant therapies in the eCRF.
9. Have received any investigational product as part of a clinical trial NOT related to the treatment of common warts within 30 days before the first application of the study drug.
10. Have epidermodysplasia verruciformis.
11. Have an active malignancy or are undergoing treatment for any malignancy.
12. Have a history or presence of clinically significant medical, psychiatric, or emotional condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the subject or the quality of the data.
13. Have a history or presence of hypersensitivity or an idiosyncratic reaction to the study drug or related compounds, or drug product excipients (acetone, ethyl alcohol, nitrocellulose, hydroxypropyl cellulose, castor oil, camphor, gentian violet, and denatonium benzoate).
14. Have a condition or situation that may interfere significantly with the subject's participation in the study (eg, subjects who required hospitalization in the 2 months before screening for an acute or chronic condition including alcohol or drug abuse), as determined by the Investigator.
15. Are sexually active or may become sexually active and are unwilling to practice a highly effective method of birth control (eg, combination of condoms and foam; oral contraceptives; intrauterine device with or without hormone release; transdermal, injectable, or intravaginal contraception). Withdrawal is not an acceptable method of birth control. Females who have reached menarche must have a negative urine pregnancy test at each visit before treatment with study drug.
16. Are pregnant or breastfeeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving complete clearance of all treatable common warts (baseline and new) at the Day 84 (EOT) Visit. | Day 84(0/+8 days)
  To evaluate the efficacy of YCANTH (VP-102) relative to Vehicle by assessing the proportion of subjects achieving complete clearance defined by complete resolution of all common warts as assessed visually by a Blinded Assessor of all treatable common warts, at the EOT Visit (Day 84).

SECONDARY OUTCOMES:
Proportion of subjects achieving sustained complete clearance of all treatable common warts (baseline and new) from Treatment Visit 4 (Day 63) through EOT Visit (Day 84). | From Day 63 (=/- 4 days) to Day 84 (0/+8 days)
  To evaluate the efficacy of YCANTH (VP-102) relative to Vehicle by assessing the proportion of subjects achieving sustained complete clearance of all treatable common warts (baseline and new) from Treatment Visit 4 (Day 63) through EOT Visit (Day 84)
Proportion of subjects achieving sustained complete clearance of all treatable common warts (baseline and new) from Treatment Visit 3 (Day 42) through EOT Visit (Day 84). | From Day 42 (+/- 4 days) to Day 84 (0/+8 days)
  To evaluate the efficacy of YCANTH (VP-102) relative to Vehicle by assessing the proportion of subjects achieving sustained complete clearance of all treatable Common warts (baseline and new) from Treatment Visit 3 (Day 42) through EOT Visit (Day 84).
Proportion of subjects achieving sustained complete clearance of all treatable common warts (baseline and new) from Treatment Visit 2 (Day 21) through EOT Visit (Day 84). | From Day 21 (+/- 4 days) to Day 84 (0/+8 days)
  To evaluate the efficacy of YCANTH (VP-102) relative to Vehicle by assessing the proportion of subjects achieving sustained complete clearance of all treatable Common warts (baseline and new) from Treatment Visit 2 (Day 21) through EOT Visit (Day 84).
Incidence and severity of AEs (including LSRs) Change from baseline in vital signs (body temperature, pulse rate). Concomitant medication use. | From enrollment to the end of Study (12 weeks to 21 weeks)
  To assess the safety of YCANTH (VP-102) relative to Vehicle, by assessing concomitant medication use and AEs (AEs), including expected LSRs.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Florida Center for Dermatology, P.A., Saint Augustine, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Anne Arundel Dermatology, PA dba Maryland Dermatology Laser Skin & Vein, Hunt Valley, Maryland
  - Tennessee Clinical Research Center, Inc., Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No